CLINICAL TRIAL: NCT05505747
Title: Enhancing Recovery Through a Combined Mechanobiologic Intervention Following Meniscus Repair
Status: Withdrawn | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Funding not awarded
Sponsor: Austin V Stone (Other)
Responsible Party: Sponsor-Investigator, Austin V Stone, Assistant Professor, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 80414
Record Dates: First submitted 2022-08-16; First posted 2022-08-18 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-05

CONDITIONS: Meniscus Tear; Meniscus; Derangement; Meniscus Lesion; Meniscus Disorder
MeSH Terms: interventions — fisetin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The study pharmacist that prepared the randomization schedule will meet with the pre-specified unblinded study personnel prior to the site initiation visit. The unblinded personnel will then prepare sealed envelopes that contain each subject's group assignment.
  The investigators will designate, a priori, study personnel that will be unblinded. These unblinded personnel will be directly involved with maintaining the drug log and communicating with participants to schedule physical therapy sessions. The unblinded pharmacist/coordinator will access the actual treatment assignment but both blinded study personnel and the patient will not know the patient's treatment assignment. The Investigator, participant, patient assessors, laboratory personnel, and statistician will remain blinded throughout the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Fisetin (Experimental): Subjects assigned to the experimental group will take approximately 20 mg/kg/day of fisetin for 2 consecutive days, followed by a 28-day senescence washout period, and then another 2-day administration. Fisetin treatment begins at 8 weeks after surgery.
  Interventions: Drug: Fisetin
- Placebo (Placebo Comparator): Subjects assigned to the experimental group will take approximately 20 mg/kg/day of placebo (corn starch) for 2 consecutive days, followed by a 28-day washout period, and then another 2-day administration. Placebo treatment begins at 8 weeks after surgery.
  Interventions: Drug: Placebo oral capsule

INTERVENTIONS:
Drug: Fisetin — Fisetin is a plant flavanol senolytic found in strawberries, persimmons, and cucumbers. This naturally derived senolytic has few side effects and previous animal models of both osteoarthritis and rheumatoid arthritis have demonstrated that the senolytic supplement fisetin reduces inflammation and slows cartilage breakdown.
  Other Names: Novusetin; 7,3',4'-flavon-3-ol; 3,3',4',7-tetrahydroxyflavone
  Arms: Fisetin
Drug: Placebo oral capsule — The oral placebo will consist of corn starch and gelatin capsules
  Arms: Placebo

SUMMARY:
Arthroscopic meniscal procedures are the most commonly performed orthopaedic procedure in the U.S. affecting 15% of Americans ages 10-65 years. Meniscus injury is also known to increase the risk of posttraumatic osteoarthritis (PTOA). The current randomized clinical trial will test a novel intervention after meniscal repair that combines an oral senolytic fisetin and real-time biofeedback program to restore joint loading and subsequent return to activity.

DETAILED DESCRIPTION:
Arthroscopic meniscal procedures are the most commonly performed orthopaedic procedure in the U.S. affecting 15% of Americans ages 10-65 years. Meniscus injury is also known to increase the risk of posttraumatic osteoarthritis (PTOA). The current randomized clinical trial will test a novel mechanobiologic intervention after meniscal repair that combines an oral senolytic fisetin and real-time biofeedback program to restore joint loading and subsequent return to activity. The premise for this program is derived from growing evidence that under-loading early after an orthopedic surgery is a major contributing factor to future PTOA development. Despite the need to assess how much force the patient can produce in various exercises to better inform progression and progress, clinicians still have few tools. By providing the realtime feedback during all exercises, the program will promote the recovery of muscle function as well which is critical for normal joint loading.

The study will 1) evaluate the feasibility and acceptability of the mechanobiologic intervention following arthroscopic repair of meniscus tears, 2) determine if the mechanobiologic intervention improves physical function, patient reported outcomes, loading and muscle strength, and biomechanical symmetry in comparison to standard of care physical therapy and oral placebo, and 3) compare cartilage composition at 1 year after meniscus surgery between the mechnobiologic intervention and a control group treated standard of care physical therapy and oral placebo.

ELIGIBILITY:
Inclusion Criteria:

Subjects will be included if all the following criteria are met:

1. Are male or female, ages 18-45;
2. Are willing to comply with all study related procedures and assessments;
3. Are ambulatory as defined by ability to complete functional performance testing;
4. Medial, lateral or combined meniscus tear treated with surgical repair.
5. Stable dose of screening/baseline medications for at least 2 months prior to the anticipated date of study drug dosing.

Exclusion Criteria:

Subjects will be excluded if any of the following criteria are met:

1. Females who are nursing, pregnant or planning to become pregnant during the duration of study drug dosing;
2. Males who do not wish to abstain from sex or use contraceptive protection during study drug dosing and for 2 weeks after the last dose;
3. Subjects who do not have the capacity to consent themselves;
4. Subjects who are unable to tolerate oral medication;
5. Subjects having previously undergone any of the following treatments in the stated time window.

   * Surgery on the Study Knee in the past 6 months;
   * Partial or complete joint replacement in the study knee. Partial or complete joint replacement in the contralateral knee is acceptable as long as the surgery was performed at least 6 months prior to enrollment and the operative knee is asymptomatic;
   * Patients who have undergone arthroscopic surgery (including microfracture and meniscectomy) on the Study Knee in the last 2 years prior to the Screening visit.
   * Patients will be excluded from the study if an Outerbridge grade III or IV chondral lesion is identified during arthroscopy.
6. Radiographic osteoarthritis (Kellgren-Lawrence Grade 2-4), full thickness chondral defect on MRI, BMI > 35 kg/m2, concomitant ligament injury, or prior ipsilateral knee ligament or meniscus surgery within prior 12 months of enrollment.
7. The following intraarticular injections:

   * Glucocorticoid within the last 2 months,
   * Extended-release corticosteroid, hyaluronic acid, or other biologic injection (platelet-rich plasma, bone marrow, adipose tissue/cells) into the Study Knee in the past 6 months within the past 6 months
   * Subjects with any of the following drug/medication statuses:
   * Currently taking Losartan;
   * Currently taking Warfarin or related anticoagulants;
   * Opioid analgesics taken in the past 8 weeks;
   * Senolytic agents taken within the past 6 months and are not willing to discontinue these medications through the duration of the study, including: Fisetin, Quercetin, Luteolin, Dasatinib, Piperlongumine, or Navitoclax;
   * Drugs that induce significant cellular stress and are not willing to discontinue these medications through the duration of the study, including alkylating agents, anthracyclines, platins, other chemotherapy drugs;
   * Medications that are sensitive substrates or substrates with a narrow therapeutic range for CYP1A2, CYP2C8, CYP2C9, CYP2C19, CYP2D6, CYP3A4, OATP1B1 or strong inhibitors or inducers of CYP3A4 (e.g. cyclosporine, tacrolimus or sirolimus);
   * Subjects taking the following other drugs if they cannot be held (per the Principal Investigator) for at least 2 days before and during administration of Fisetin: cyclosporine, tacrolimus, repaglinide, and bosentan.
   * Subjects with any of the following disease statuses:
   * Significant liver disease (i.e. greater than or equal to 2x the upper limit of normal bilirubin levels) or as in the opinion of the Principal Investigator;
   * Significant renal disease (eGFR of <60 ml/min/1.73m2) or as in the opinion of the Principal Investigator;
   * History of other formally diagnosed joint diseases including osteonecrosis, acromegaly, Paget's disease, Ehlers-Danlos Syndrome, Gaucher's disease, Cushing's syndrome, Stickler's syndrome, joint infection, hemophilia, hemochromatosis, or neuropathic arthropathy of any cause;
   * Any active systemic autoimmune disease with musculoskeletal involvement or any history of system inflammatory arthritis;
   * Patients with type 1 or 2 diabetes (HbA1c>6.5%) and/or taking medications that affect insulin levels, including: Metformin (within the last week), Glucocorticoids (within the last month), Acarbose (within the last week);

9. Those with moderate to severe depression (PHQ-9 score > 10) will also be excluded since knee OA patients with depression have previously demonstrated worse pain trajectories; 10. Subjects that have any medical condition, including laboratory findings and findings in the medical history or in the pre-study assessments, that in the opinion of the Investigator constitutes a risk or contraindication for participation in the study or that could interfere with the study objectives, conduct or evaluation or prevent the patient from fully participating in all aspects of the study.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2025-07 (Estimated); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Change in International Knee Documentation Committee (IKDC) Score between baseline and 1 year | Baseline, 1 year
  The IKDC Score was designed to assess patients with a variety of knee disorders including meniscal injuries. The IKDC consists of 18 items, and scores range from 0 points (lowest level of function or highest level of symptoms) to 100 points (highest level of function and lowest level of symptoms).

SECONDARY OUTCOMES:
Change in MRI T1rho between baseline and 1 year | Baseline, 1 year
  Increased T1rho relaxation times have been associated with loss of proteoglycan content. This then corresponds with MRI changes associated with the loss of proteoglycan content.

CONTACTS AND LOCATIONS:
Overall Officials: Austin Stone, MD, PhD, Principal Investigator — University of Kentucky
Locations (1):
- UK Healthcare at Turfland, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No